CLINICAL TRIAL: NCT02912689
Title: Non-invasive Ventilation (NIV) - Neurally Adjusted Ventilatory Assist (NAVA) vs NIV for Acute Hypercapneic Respiratory Failure in COPD: A Randomized Controlled Trial
Brief Title: NIV - NAVA vs NIV - PS for COPD Exacerbation
Acronym: NAVA-NICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Vijay Hadda, Assistant Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IECPG/360/29.06.2016
Record Dates: First submitted 2016-09-04; First posted 2016-09-23 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: COPD Exacerbation
Keywords: COPD; Non-invasive ventilation; NAVA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurally adjusted ventilator assist (Experimental): Neurally adjusted ventilator assist (NAVA) during NIV for exacerbation of COPD.
  Interventions: Device: Neurally Adjusted Ventilator Assist
- Pressure support ventilation (Active Comparator): Pressure support ventilation (PSV) during NIV for exacerbation of COPD.
  Interventions: Device: Pressure support ventilation

INTERVENTIONS:
Device: Neurally Adjusted Ventilator Assist — NAVA during Non-invasive ventilation
  Other Names: NAVA
  Arms: Neurally adjusted ventilator assist
Device: Pressure support ventilation — PS during Non-invasive ventilation
  Other Names: PSV
  Arms: Pressure support ventilation

SUMMARY:
Number of Patients:

Total no. of patients = 40 patients NIV-PSV group (Group A) = 20 NIV-NAVA group (Group B) = 20

Inclusion criteria

a) Patients of Chronic obstructive pulmonary disease with acute hypercapnic respiratory failure (pH < 7.35 and PaCO2 >45 mmHg) requiring noninvasive ventilation and with no indication for invasive mechanical ventilation.

Exclusion criteria

1. Patient with any contra-indication for insertion of nasogastric tube (like recent gastrointestinal bleeding in previous 30 days, esophageal varices)
2. Patient with any contraindication of noninvasive ventilation (such as hemodynamic instability, active gastrointestinal bleed etc)
3. Patients with a known neuromuscular, central or peripheral nervous system disorder.
4. Patient not willing to give consent.

Control(s): Patients receiving pressure support ventilation (NIV-PSV) will act as control

Study design: Randomized interventional study

Dosages of drug: None

Duration of treatment: Till patient improves or requires invasive ventilation.

Brief Methodology Patients of COPD with acute exacerbation will be randomized into two groups (group A and group B) to receive NIV-PSV or NIV-NAVA respectively. A special naso-gastric catheter (EAdi-catheter) will be placed in all patients. In each mode, NIV will be applied using a non-vented oro-nasal mask that will be fitted enough to avoid air leaks. Patients in Group A will receive NIV-PS and Group B will receive ventilation via NIV-NAVA. Pressure support and PEEP levels will be set by the treating physician to achieve a tidal volume (Vt) of 6 to 8 mL/kg of ideal body weight. NAVA level will be adjusted to match peak pressures of NIV-PSV using manufacturer-supplied software. After stabilization, a 30-min period of each NIV trial will be recorded and manually analyzed offline. Subsequent readings will be taken at 2, 6 and at 24 hours and then at 6 hourly interval from day 2 onwards. In each trial, patient-ventilator asynchronies (ineffective efforts, auto triggering, premature cycling, delayed cycling, and double triggering) will be determined on EAdi, airway pressure, and flow signal. The number of each type of asynchrony, defined as the number of events per minute, will be determined for each recording period. The asynchrony index (AI), in percentage, will be calculated as described previously, and an AI >10% will be considered severe asynchrony. Patient comfort level after each mode of ventilation will be assessed by using visual analogue scale. Various clinical, ventilatory and arterial blood gas parameters will be recorded.

Statistical analysis Data will be expressed as mean ± standard deviation (SD), or percentage. Differences in continuous variables between the two groups will be compared using student's t test (or Mann-Whitney U test); while differences in categorical data will be compared using the chi- square test (or Fisher's exact test). A p value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Chronic obstructive pulmonary disease with acute hypercapnic respiratory failure requiring noninvasive ventilation and with no indication for invasive mechanical ventilation will be included in the study.

Exclusion Criteria:

* Patient with any contraindication for insertion of nasogastric tube (like recent gastrointestinal bleeding in previous 30 days, Esophageal varices)
* Patient with any established contraindication of noninvasive ventilation. (Like Hemodynamic instability, active GI bleed etc)
* Patients with a known neuromuscular, Central or peripheral nervous system disorder.
* Patient not willing to give consent.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in the number of patient ventilator asynchrony | Entire period of ventilatory support, an average of 5 days
  To assess the difference of number of patient ventilator asynchrony

SECONDARY OUTCOMES:
Difference in rate of NIV failure | Entire hospital stay, an average of 7 days
  To assess the difference of rate of NIV failure
Difference in total duration of ventilatory support | Entire hospital stay, an average of 7 days
  To assess the difference in total duration of ventilatory support

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Hadda, MD, Principal Investigator — AIIMS, New Delhi, INDIA
Locations (1):
- AIIMS, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Will share, if required

REFERENCES:
- [Derived] Tajamul S, Hadda V, Madan K, Tiwari P, Mittal S, Khan MA, Mohan A, Guleria R. Neurally-Adjusted Ventilatory Assist Versus Noninvasive Pressure Support Ventilation in COPD Exacerbation: The NAVA-NICE Trial. Respir Care. 2020 Jan;65(1):53-61. doi: 10.4187/respcare.07122. Epub 2019 Oct 22. PMID 31641071